CLINICAL TRIAL: NCT04441918
Title: A Randomized, Double-blind, Placebo-controlled, Phase I Clinical Study to Evaluate the Tolerability, Safety, Pharmacokinetic Profile and Immunogenicity of JS016 (Anti-SARS-CoV-2 Monoclonal Antibody) Injection in Chinese Healthy Subjects After Intravenous Infusion of Single Dose
Brief Title: Tolerability,Safety,Pharmacokinetic Profile and Immunogenicity of a Recombinant Humanized Anti-SARS-CoV-2 Monoclonal Antibody (JS016) for Injection in Chinese Health Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JS016-001-I
Record Dates: First submitted 2020-06-06; First posted 2020-06-22 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: COVID-19; and High Infection Risk of SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — etesevimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental)
  Interventions: Combination Product: JS016 (anti-SARS-CoV-2 monoclonal antibody)
- Control group (Experimental)
  Interventions: Combination Product: JS016 (anti-SARS-CoV-2 monoclonal antibody)

INTERVENTIONS:
Combination Product: JS016 (anti-SARS-CoV-2 monoclonal antibody) — JS016 (anti-SARS-CoV-2 monoclonal antibody)

SUMMARY:
This is a randomized, double-blind, placebo-controlled, phase I clinical study to evaluate the tolerability, safety, pharmacokinetic profile and immunogenicity of JS016 (anti-SARS-CoV-2 monoclonal antibody) injection in Chinese healthy subjects after intravenous infusion of single dose.Eligible patients will be injection JS016 (anti-SARS-CoV-2 monoclonal antibody)

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged 18 to 45 years, inclusive;
2. The body weight no less than 50 kg for male subjects and no less than 45 kg for female subjects. Body mass index (BMI) = weight (kg)/square of height (m2), ranging from 18-28 kg/m2 (including the critical value);
3. Normal or abnormal but clinically insignificant physical examination, vital signs, laboratory tests and other accessory examinations (chest radiology, abdominal B-mode ultrasonography, ECG, etc.);
4. No plan of pregnancy and being willing to use effective contraceptive measures for subject (including partner) from informed consent to 6 months after administration of investigational product, see Appendix 5 for the specific contraceptive measures;
5. The subjects are able to understand the content of the study and voluntary to sign the informed consent form; meanwhile, being able to complete the study as required in the protocol.

Exclusion Criteria:

Excluded for novel coronavirus (SARS-CoV-2) infection

1. Having one of the following evidence on SARS-CoV-2 infection:

   1. SARS-CoV-2 determined by reverse transcription-polymerase chain reaction (RT-PCR) and/or next generation sequencing (NGS) in diagnostic specimens (nasopharyngeal swabs) during screening and pre-randomization (results within 3 days before randomization are accepted);
   2. Previous viral gene sequencing showed high homology with the known SARS-CoV-2;
   3. Positive specific antibody IgM or IgG against serum SARS-CoV-2; Excluded for previous and concomitant medications
2. Previous vaccination of SARS-CoV-2 vaccine or having participated in the clinical trial on SARS-CoV-2 neutralizing antibody;
3. Use of therapeutic biologics within 12 weeks prior to screening, or remaining in the elimination period of the drug (within 5 half-lives) at random administration, whichever is longer;
4. Participation in any other clinical study with intervention of investigational product within 4 weeks prior to screening, or remaining in the elimination period of the drug (within 5 half-lives) prior to screening, whichever is longer;
5. Vaccination of vaccine within 12 weeks prior to screening, or plan to use Bacille Calmette-Guérin vaccine or other vaccine during the study and within 12 weeks after the study;
6. Use of hydroxychloroquine, herbal medicine, any prescription drug or over-the-counter drug within (inclusive) 14 days prior to screening; Surgery
7. Any major surgery within 8 weeks (inclusive) prior to screening, or requiring such surgery during the study, and such surgery is considered by the investigator to possibly bring unacceptable risk for subjects upon confirmation with the sponsor; Abnormal physical examination, laboratory examination and history
8. Lying systolic blood pressure (SBP) > 140 mmHg or < 90 mmHg, and/or diastolic blood pressure (DBP) > 90 mmHg or < 50 mmHg at screening and randomization;
9. Total white blood cell (WBC) count < 3.5 x 109/L, platelet < 140 x 109/L, neutrophil < 2.0 x 109/L, or hemoglobin decreased (male < 135 g/L, female < 120 g/L), lymphocytes < 1.0 x 109/L at screening;
10. ALT or AST > 2 × upper limit of normal, or eGFR ≤ 90 mL/min/1.73m2 at screening;
11. Abnormal ECG at screening, single QTcF > 450 msec, and/or other abnormalities of clinical significance, unacceptable risk that may be brought by participation in the study;
12. History of HIV infection, and/or positive aiti-HIV antibody, positive hepatitis B surface antigen (HBsAg), positive hepatitis C antibody (anti-HCV), or positivetreponema pallidum particle agglutination test (TPPA) at screening;
13. History of transplantation of vital organs (e.g., heart, lung, liver, kidney, etc.);
14. Having malignant tumor (excluding the malignant tumor cured with no recurrence in the past 5 years, completely resected basal cell and squamous cell carcinoma of skin, completely resected carcinoma in situ of any type);
15. Other major diseases within one year;
16. Medical history and previous history suggest the following diseases: including but not limited to gastrointestinal, renal, hepatic, neurological, hematological, endocrine, oncological, pulmonary, immune, mental or cerebro- and cardiovascular diseases; Substance abuse, alcohol abuse
17. History of drug abuse or use of narcotics in the past 5 years, or positive urine drug screening;
18. History of alcohol abuse or intake of excessive alcohol in the past 6 months (14 units of alcohol per week: 1 unit = 285 mL beer, or 25 mL liquor, or 100 mL wine), or alcohol test positive; History of allergies
19. Known serious allergic reaction or hypersensitive to food, inhaled and contact material as well as drugs, or allergic constitution (allergy to various drugs and food);
20. Known history of allergy or hypersensitivity to the investigational drug, other monoclonal antibody drugs and therapeutic protein preparations (fresh or frozen plasma, human serum albumin, cytokine, interleukin etc.); Pregnancy, lactation
21. Positive β-Human Chorionic Gonadotropin (β-HCG) or breastfeeding female subjects; Blood loss and others
22. Subjects who lost blood or donated more than 400 mL, or received blood transfusion in the past 3 months; or plan to donate blood during the study;
23. Any other condition that the subject is considered by the investigator as inappropriate to participate in the study, for example, potential compliance issue, inability to complete all the tests and evaluations according to the requirements in the protocol, or uncontrolled mental, neurological or psychological disorders, participation in the study is judged by the investigator to be associated with uncontrollable risk.

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-06-05 (Actual); Primary Completion 2020-12-11 (Estimated); Study Completion 2020-12-11 (Estimated)

PRIMARY OUTCOMES:
Correlation of adverse events with the investigational product | 12 Weeks
  Any adverse event, serious adverse event (SAE) occurred during the clinical study, including clinical symptoms and abnormal vital signs, abnormal laboratory tests (complete blood cell count, serum chemistry, routine urinalysis, coagulation function, etc.) and 12-lead ECGs will be observed for all the subjects, the their clinical manifestations and features, severity, time to onset, end time, therapeutic measures and outcomes will be recorded, and the correlation of the adverse events with the investigational product will be judged

SECONDARY OUTCOMES:
Primary pharmacokinetic variables | 12 Weeks
  Area under the curve from the time of dosing to the last measurable concentration time t (AUC0-last);
Primary pharmacokinetic variables | 12 Weeks
  Maximum concentration (Cmax);
Primary pharmacokinetic variables | 12 Weeks
  Mean residence time (MRT)
Primary pharmacokinetic variables | 12 Weeks
  Terminal half life (t1/2);

OTHER OUTCOMES:
pharmacokinetic | 12 Weeks
  Area under the analyte concentration-time curve from time 0 and extrapolated to infinite time (AUC0-∞);
pharmacokinetic | 12 Weeks
  Time to maximum concentration (Tmax);
pharmacokinetic | 12 Weeks
  Clearance (CL);
pharmacokinetic | 12 Weeks
  Apparent terminal elimination rate constant (λz)
pharmacokinetic | 12 Weeks
  Apparent volume of distribution (Vd)

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital affiliated to Fudan University, Shanghai, China

REFERENCES:
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343
- [Derived] Wu X, Li N, Wang G, Liu W, Yu J, Cao G, Wang J, Chen Y, Ma J, Wu J, Yang H, Mao X, He J, Yu Y, Qiu C, Li N, Yao S, Feng H, Yan J, Zhang W, Zhang J. Tolerability, Safety, Pharmacokinetics, and Immunogenicity of a Novel SARS-CoV-2 Neutralizing Antibody, Etesevimab, in Chinese Healthy Adults: a Randomized, Double-Blind, Placebo-Controlled, First-in-Human Phase 1 Study. Antimicrob Agents Chemother. 2021 Jul 16;65(8):e0035021. doi: 10.1128/AAC.00350-21. Epub 2021 Jul 16. PMID 33972256